CLINICAL TRIAL: NCT05535101
Title: Exploration of Non-invasive Theta Burst Stimulation in Patients With Methamphetamine Use Disorder: Efficacy and Mechanism
Brief Title: Non-invasive Brain Stimulation in Patients With Methamphetamine Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111-019-F
Record Dates: First submitted 2022-04-27; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-04

CONDITIONS: Craving; Depression, Anxiety; Amphetamine Addiction
Keywords: Addiction; amphetamine; non-invasive theta burst stimulation
MeSH Terms: conditions — Depression; Anxiety Disorders; Amphetamine-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- theta burst stimulation (Experimental): Those participants to receive 1-3 sessions in a single day at an interval of 15 minutes(at least), and 5 high-frequency iTBS sessions per week in total four weeks. Each session: 600-900 pulses with 120-100% resting motor threshold.
  Interventions: Device: Intermittent theta burst transcranial magnetic stimulation (iTBS)
- Sham arm (Sham Comparator): Sham stimulation was delivered using the same protocol as active stimulation, but with the TMS coil rotated by 90 degrees with the edge of the coil touching the scalp.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Intermittent theta burst transcranial magnetic stimulation (iTBS) — The amphetamine users will undergo a one-month iTBS intervention. From Week 1 to Week 4, subjects will be treated five times a week.
  Arms: theta burst stimulation
Device: Sham stimulation — Sham stimulation was delivered using the same protocol as active stimulation, but with the TMS coil rotated by 90 degrees with the edge of the coil touching the scalp.
  Arms: Sham arm

SUMMARY:
The study aims to apply the intermittent theta burst transcranial magnetic stimulation (iTBS) treatment and evaluate the effect in improving craving, affective symptoms, and cognitive function for those participants in the community with amphetamine use. An electroencephalography and blood biomarkers will also be examined to explore the possible mechanisms.

DETAILED DESCRIPTION:
In this study, participants with amphetamine use will be recruited from psychiatric clinics. They will be randomly assigned to two different transcranial magnetic stimulation groups, the iTBS and sham groups. Those participants to receive 1-3 sessions in a single day at an interval of 15 minutes, and 5 high-frequency iTBS sessions per week in total four weeks. After the completion of the four-week course, the severity of symptoms for the next one month and three months will be tracked.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged 20-65.
2. Diagnosis as amphetamine use disorder by clinical psychiatrist according to DSM-V

Exclusion Criteria:

1. Major disorders other than substance use disorders in Diagnostic and Statistics Manual-5 (e.g. Schizophrenia, organic brain syndrome, and bipolar disorders).
2. Epilepsy, head trauma, migraine, cardiovascular comorbidity, atypical parkinsonian disorder
3. patients with heart pacemakers, implanted drug delivery aids, artificial electronic ears, implantable defibrillators, and/or implanted nerve stimulators, and near the implants mentioned above.
4. patients with metal implants above the chest.
5. people who have damaged skin in areas of the patient's body that receive stimulation.
6. patients with multiple sclerosis.
7. patients who have extensive ischemic scarring.
8. pregnant women.
9. patients with a family history of spasms/epilepsy
10. patients taking medications that may lower the seizure threshold.
11. patients with severe sleep disorders related to previous rTMS treatment.
12. patients with severe heart disease
13. patients with intracranial stress caused by uncontrollable migraines.
14. people who have been evaluated by a physician as unfit to participate in clinical trials.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (Taiwanese version) | Baseline(Week 0, before intervention), Week 4(after iTBS program), Week 8, Week 16
  Respondents will specify their level of craving from none to extreme on a 100 mm line (score: 0-10) in each questionnaires, and there are nine questionnaires related to craving.

SECONDARY OUTCOMES:
The Beck depression inventory (Taiwanese version BDI) | Baseline(Week 0, before intervention), Week 4(after iTBS program), Week 8, Week 16
  The Beck depression inventory (Taiwanese version BDI) will be applied to evaluate the depression during the period of methamphetamine abstinence. (Total score: 0-63)
The Beck anxiety inventory (Taiwanese version BAI) | Baseline(Week 0, before intervention), Week 4(after iTBS program), Week 8, Week 16
  The Beck anxiety inventory (Taiwanese version BAI) will be applied to evaluate the anxiety during the period of methamphetamine abstinence. (Total score: 0-63)
Cognitive function | Baseline(Week 0, before intervention), Week 4(after iTBS program), Week 8, Week 16
  Continuous performance test was developed by Rosvold and designed as a computerized test of cognitive function.The outputs include hit rates, correct percentages, and answer time for each item. Generally, higher correct percentage with shorter answer time mean better attention.
Tolerance | Post intervention everytime (8 times total)
  The respondents will specify five physical symptoms which might related to rTMS intervention (Yes/No: headache, local pain/discomfort, head/face pain/discomfort, seizure, hearing loss/ear ache)
blood biomarkers | Baseline(Week 0, before intervention), Week 4(after iTBS program), Week 8, Week 16
  Three biomarker reflecting neuron inflammation or neuron damage will be measured using blood samples, including C-C Motif chemokine ligand 11, neurofilament light chain and exosomal RNA to explore the possible mechanism of iTBS.
Electroencephalography | Baseline(Week 0), Week 4
  The EEG will be perform to collect the parameters across broad brain regions to transform into subsequent information of functional connectivity, including phase locking value (PLV) across all electrodes for delta, theta, alpha, and beta frequency bands.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Che Chen, MD, MSc, Principal Investigator — Physician, Department if Psychiatry, National Taiwan University Hospital Hsin-Chu branch